CLINICAL TRIAL: NCT01288638
Title: A Lifestyle Intervention for Women With Polycystic Ovary Syndrome: The Role of a Pulse-Based Diet and Aerobic Exercise on Infertility Measures and Metabolic Syndrome Risk
Brief Title: Lifestyle Intervention for Polycystic Ovary Syndrome: Pulse-Based Diet and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Saskatchewan Pulse Growers (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pulse-PCOS
Record Dates: First submitted 2011-01-13; First posted 2011-02-02 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Polycystic Ovary Syndrome; Metabolic Syndrome
Keywords: Polycystic Ovary Syndrome; Metabolic Syndrome; Pulse; Lifestyle Intervention; Aerobic Exercise; Diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulse-based diet (Experimental): The pulse based-diet will include meals prepared with dry peas, lentils, chickpeas, and beans. Two meals will be supplied daily for 16 weeks to those participants on the pulse-based diet program. Meals will contain approximately 90g dried peas, 225 g chickpeas or beans, or 150g lentils.
  Interventions: Other: Pulse-based diet
- TLC diet (Placebo Comparator): Grocery gift cards will be provided weekly for 16 weeks to those participants in the placebo group. Recipe booklet will be given to follow Therapeutic Lifestyle Changes (TLC) guidelines, recommended by National Cholesterol Education Program (NCEP) and will be based on lean-meats for the protein source. The recipes will exclude pulses.
  Interventions: Other: TLC diet

INTERVENTIONS:
Other: Pulse-based diet — The pulse based-diet will include meals prepared with dry peas, lentils, chickpeas, and beans. Two meals will be supplied daily for 16 weeks to those participants on the pulse-based diet program. Meals will contain approximately 90g dried peas, 225 g chickpeas or beans, or 150g lentils.
  Arms: Pulse-based diet
Other: TLC diet — Grocery gift cards will be provided weekly for 16 weeks to those participants in the placebo group. Recipe booklet will be given to follow Therapeutic Lifestyle Changes (TLC) guidelines, recommended by National Cholesterol Education Program (NCEP) and will be based on lean-meats for the protein source. The recipes will exclude pulses.
  Arms: TLC diet

SUMMARY:
The purpose of our study is to evaluate the effectiveness of a lifestyle program for women with Polycystic Ovary Syndrome (PCOS). The investigators want to assess the effect of a pulse-based diet (i.e. a diet that contains lentils, chick-peas, peas, and beans) and aerobic exercise for improving PCOS disease features and risk factors for metabolic syndrome. We would like to determine the therapeutic effects of a lifestyle program that combines a pulse-based diet and exercise on the multiple disease measures of PCOS and metabolic syndrome.

DETAILED DESCRIPTION:
To date, we have developed the pulse-based and meat-based healthy meals following Therapeutic Lifestyle Changes (TLC)guidelines recommended by NCEP for the intervention. We have been recruiting and enrolling participants into the study with our few set of participants having completed the 4 month intervention. Baseline data have been also collected on all participants assessed for PCOS. Preliminary measurements on POCS characteristics, baseline dietary and exercise habits of women with PCOS will be soon available.

This study involves an intervention comparing a diet containing pulses (i.e. beans, peas, chick peas, lentils) to a diet recommended by the National Cholesterol Education Program (NCEP) for improving markers of metabolic syndrome and fertility in women with poly cystic ovarian syndrome who are also enrolled in an aerobic exercise program. To date, seven women in the pulse-diet group have completed the intervention, nine women in the group receiving the NCEP diet have completed the intervention, four women are currently enrolled on the pulse diet and two women are currently enrolled on the NCEP diet.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of PCOS
* Aged 18-35 years

Exclusion Criteria:

* Taking birth control or fertility medications
* Medical conditions that limit exercise or which limit consumption of a pulse-based diet (allergies or intolerances)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2011-01; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in polycystic ovary syndrome disease measures from baseline | At baseline, before TLC lead-in, twice during the intervention, at 6 months follow-up and at 12 months follow-up

SECONDARY OUTCOMES:
Change in metabolic syndrome disease measures from baseline | At baseline, before TLC lead-in, twice during the intervention, at 6 months follow-up and at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gordon A Zello, PhD, Principal Investigator — University of Saskatchewan; Philip Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] McBreairty LE, Chilibeck PD, Chizen DR, Pierson RA, Tumback L, Sherar LB, Zello GA. The role of a pulse-based diet on infertility measures and metabolic syndrome risk: protocol of a randomized clinical trial in women with polycystic ovary syndrome. BMC Nutr. 2017 Mar 7;3:23. doi: 10.1186/s40795-017-0142-6. eCollection 2017. PMID 32153805
- [Derived] Kazemi M, Pierson RA, McBreairty LE, Chilibeck PD, Zello GA, Chizen DR. A randomized controlled trial of a lifestyle intervention with longitudinal follow-up on ovarian dysmorphology in women with polycystic ovary syndrome. Clin Endocrinol (Oxf). 2020 Jun;92(6):525-535. doi: 10.1111/cen.14179. Epub 2020 Mar 16. PMID 32092167
- [Derived] Kazemi M, McBreairty LE, Zello GA, Pierson RA, Gordon JJ, Serrao SB, Chilibeck PD, Chizen DR. A pulse-based diet and the Therapeutic Lifestyle Changes diet in combination with health counseling and exercise improve health-related quality of life in women with polycystic ovary syndrome: secondary analysis of a randomized controlled trial. J Psychosom Obstet Gynaecol. 2020 Jun;41(2):144-153. doi: 10.1080/0167482X.2019.1666820. Epub 2019 Sep 27. PMID 31558086
- [Derived] Kazemi M, McBreairty LE, Chizen DR, Pierson RA, Chilibeck PD, Zello GA. A Comparison of a Pulse-Based Diet and the Therapeutic Lifestyle Changes Diet in Combination with Exercise and Health Counselling on the Cardio-Metabolic Risk Profile in Women with Polycystic Ovary Syndrome: A Randomized Controlled Trial. Nutrients. 2018 Sep 30;10(10):1387. doi: 10.3390/nu10101387. PMID 30274344